CLINICAL TRIAL: NCT01051362
Title: Phase II Study of Pegylated Liposomal Doxorubicin and Carboplatin as First Line Treatment for Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Pegylated Liposomal Doxorubicin and Carboplatin as First Line Treatment for Patients With Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Department of Cardiothoracic Surgery, The First Affiliated Hospital of Guangzhou Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAHG20060216
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2006-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Advanced Non-small Cell Lung Cancer; Pegylated liposomal doxorubicin; Carboplatin; Chemotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 1-dodecylpyridoxal; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PLD and Carboplatin (No Intervention): Pegylated liposomal doxorubicin (PLD) 30 mg/m2, followed by Carboplatin AUC (area under the curve) 5, every 21 days for 4 cycles or until progression.
  Interventions: Drug: PLD and Carboplatin

INTERVENTIONS:
Drug: PLD and Carboplatin — Pegylated liposomal doxorubicin (PLD) 30 mg/m2, followed by Carboplatin AUC (area under the curve) 5, every 21 days for 4 cycles or until progression.

SUMMARY:
This Phase II study is to explore the efficacy and toxicity of Pegylated liposomal doxorubicin and Carboplatin in patients with previously untreated non-small cell lung cancer (NSCLC) not amenable to radiotherapy or surgical treatment. The planned enrollment for this trial is 48 patients (including a 10% rate for inevaluable patients).

DETAILED DESCRIPTION:
Pegylated liposomal doxorubicin (PLD) is the first antineoplastic drug derived from the new technology of liposome formulation to be introduced in clinical practice. The low myocardium uptake of this formulation accounts for its reduced cardiac toxicity, confirmed both in preclinical models and in humans. Preclinical data have shown activity in NSCLC xenografts. This Phase II study is to explore the efficacy and toxicity of Pegylated liposomal doxorubicin and Carboplatin in patients with previously untreated non-small cell lung cancer (NSCLC) not amenable to radiotherapy or surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small-cell bronchogenic carcinoma (squamous carcinoma, adenocarcinoma, or large cell carcinoma). Cytologic specimens obtained by brushings, washings, or needle aspiration of the defined lesion are acceptable. Mixed tumors with small-cell anaplastic elements are not eligible.
* Patients who have newly diagnosed unresectable stage III or IV disease are eligible. Patients with stage III disease should be ineligible for combined modality therapy (i.e., pleural effusions, pericardial effusions, etc.).
* Patients must not have received any prior antineoplastic chemotherapy for metastatic lung cancer prior to study entry.
* Patients who have had previous radiotherapy as definitive therapy for locally advanced non-small-cell are eligible as long as the recurrence is outside the original radiation port. Radiation therapy must have been completed greater than 4 weeks prior to registration.
* Male or female patients >=18 years of age.
* Life expectancy of at least 3 months.
* ECOG performance status of <=2.
* Measurable disease by RECIST criteria.
* Laboratory values as follows: ANC >=1500/mm3 (7 days prior to treatment); Hemoglobin >=8 g/dL;Platelets >=100,000 mm3 (7 days prior to treatment); Bilirubin <=1 x ULN for institution; AST/SGOT <=2.5 x ULN or <=5.0 x ULN in patients with liver metastases and ALT/SGPT <=2.5 x ULN or <=5.0 x ULN in patients with liver metastases; Creatinine <=2.0 mg/dL or Calculated (measured) GFR >=40 mL/min; PT/INR and PTT <=1.5 x ULN
* Peripheral neuropathy <= grade 1.
* Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment.
* Patient must be accessible for treatment and follow-up.
* All patients must be able to understand the nature of the study and give written informed consent prior to study entry.

Exclusion Criteria:

* A history of cardiac disease as defined by malignant hypertension, unstable angina, congestive heart failure of > grade 2 per New York Heart Association (NYHA) criteria, myocardial infarction within the previous 6 months, or symptomatic cardiac arrhythmias.
* Metastatic brain or meningeal tumors.
* Uncontrolled intercurrent illness.
* Chemotherapy, investigational drug therapy, or major surgery ≤ 4 weeks prior to starting study drug, or patients who have not recovered from side effects of previous therapy.
* Patient is <=5 years free of another primary malignancy, except if the other primary malignancy is not currently clinically significant or requiring active intervention, or if the other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
* Concomitant use of any anti-cancer therapy or radiation therapy.
* Other concurrent severe, uncontrolled infection or intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
To evaluate the overall response rate (complete and partial responses) in previously untreated advanced non-small-cell lung cancer (NSCLC) treated with Pegylated liposomal doxorubicin and Carboplatin | 3 months

SECONDARY OUTCOMES:
To evaluate the progression-free survival (PFS) and overall survival (OS) in previously untreated advanced NSCLC treated with Pegylated liposomal doxorubicin and Carboplatin | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, MD, FACS, Principal Investigator — Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College
Locations (1):
- Department of Cardiothoracic Surgery, the First Affiliated Hospital of Guangzhou Medical College, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Numico G, Castiglione F, Granetto C, Garrone O, Mariani G, Costanzo GD, Ciura PL, Gasco M, Ostellino O, Porcile G, Merlano M. Single-agent pegylated liposomal doxorubicin (Caelix) in chemotherapy pretreated non-small cell lung cancer patients: a pilot trial. Lung Cancer. 2002 Jan;35(1):59-64. doi: 10.1016/s0169-5002(01)00269-0. PMID 11750714